CLINICAL TRIAL: NCT06655987
Title: Effects of Unrestrained Femoral Internal Rotation Manipulation on Hip External Rotation Strength in Individuals With Nonspecific Hip Pain: A One-Week Follow-Up Clinical Trial
Brief Title: Hip Manipulation for Improved Strength in Patients With Hip Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrews University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 24-062
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hip Pain
Keywords: Hip Pain; Hip Weakness; UFIR Manipulation; Manual Therapy; Physical Therapy; Joint Manipulation; Hip External Rotation Strength

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Participants receiving the Unrestrained Femoral Internal Rotation (UFIR) manipulation.
  Interventions: Other: Unrestrained Femoral Internal Rotation (UFIR) manipulation
- Control Group (Placebo Comparator): Participants receiving a sham manipulation (gentle hand placement)
  Interventions: Other: Sham manipulation

INTERVENTIONS:
Other: Unrestrained Femoral Internal Rotation (UFIR) manipulation — This is the primary intervention applied to the experimental group. It involves a high-velocity, low-amplitude thrust at the greater trochanter of the affected hip, intended to improve joint mobility and potentially address neuromuscular dysfunction contributing to hip pain and weakness.
  Arms: Experimental Group
Other: Sham manipulation — This serves as the control intervention. It involves gentle hand placement over the affected hip's external rotators for a brief duration. This is intended to mimic the physical contact of the UFIR manipulation without actually delivering the therapeutic thrust.
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate the potential effects of an unrestrained femoral internal rotation (UFIR) manipulation technique on hip external rotation strength in individuals with nonspecific hip pain. The results of this study may help physical therapists and other healthcare professionals to better understand the effectiveness of this technique in improving hip strength and function in patients with nonspecific hip pain.

DETAILED DESCRIPTION:
Background and Rationale

Hip pain is a prevalent and debilitating condition affecting adults of all ages and activity levels, with significant impact on daily function. In athletes, the rates of hip injuries are particularly high. The heterogeneity of nonspecific hip pain, coupled with limited research on accurate diagnosis and treatment, poses challenges for physical therapists.

This study focuses on the potential of joint manipulation, particularly the Unrestrained Femoral Internal Rotation (UFIR) technique, to improve hip external rotation strength in individuals with nonspecific hip pain and weakness. While strength training is commonly used to address hip weakness, there's a lack of research on alternative approaches like joint manipulation. This research seeks to bridge this gap and explore the potential benefits of UFIR manipulation in enhancing hip function and reducing pain.

Research Procedures

Design: Prospective, randomized, controlled trial Setting: SKYE Physiotherapy, Columbia, MD Sample: 24 adults (18-55 years) with nonspecific hip pain and ipsilateral hip external rotation weakness Intervention: Experimental group receives UFIR manipulation, control group receives sham manipulation Outcome Measures: Bilateral hip external rotation strength assessed by manual muscle testing (MMT) and hand-held dynamometer (HHD) at baseline, immediately post-intervention, and 1-week follow-up.

Data Analysis: Descriptive statistics, Friedman test, Kruskal-Wallis test, ANOVA, and repeated measures ANOVA will be used to analyze data.

Study Procedures

Recruitment: Participants will be recruited through flyers and social media platforms.

Screening and Enrollment: Eligible participants will complete an electronic health screening form and provide informed consent.

Randomization: Participants will be randomly assigned to either the experimental or control group.

Intervention: The examiner will administer UFIR manipulation to the experimental group and sham manipulation to the control group.

Assessments: Hip external rotation strength will be measured using MMT and HHD at baseline, immediately post-intervention, and at 1-week follow-up.

Data Analysis: Statistical analysis will be performed to assess changes in hip external rotation strength within and between groups.

Internal Validity and Generalizability

The study acknowledges potential threats to internal validity, including testing effects, instrumental bias, and experimenter bias. Measures to mitigate these threats include standardized techniques, a one-week interval between assessments, and randomization. The study aims to recruit a diverse sample from Howard County, MD, to enhance external validity and generalizability of findings.

Conclusion

This study aims to contribute to the understanding of the potential benefits of joint manipulation, specifically UFIR, in improving hip external rotation strength and function in individuals with nonspecific hip pain and weakness. The findings may inform clinical practice and provide alternative treatment options for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* individuals who meet the following inclusion criteria will be eligible to participate in this study: 1) nonspecific hip pain, 2) ipsilateral hip external rotation weakness (at or below 3+) based on the MMT test

Exclusion Criteria:

* individuals who meet any of the following exclusion criteria will not be eligible to participate in this study: 1) do not speak English, 2) have an impaired cognition and are unable to follow multi-step commands, 3) require an assistive device for standing balance, 4) have complaints of intractable (intolerable) pain, 5) have a history of hip dislocation or total hip replacement, 6) have a history of hip fracture or arthroscopy in the past 6 months, 7) have a history of lumbar spine fracture or surgery (e.g., lumbar discectomy and fusion) in the past 6 months, 8) present with neurological condition (i.e., stroke, Parkinson's disease, or lumbar radiculopathy), 9) known congenital hip dysplasia/adolescent hip disease, and 10) known osteoporosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Change in hip external rotation strength (measured in pounds using a hand-held dynamometer) | Baseline (pre-intervention), immediately post-intervention, and one-week follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- SKYE Physiotherapy, Columbia, Maryland, United States

IPD SHARING:
Plan to Share IPD: No